CLINICAL TRIAL: NCT03946748
Title: An Open-Label, Single Arm Study to Evaluate the Efficacy and Safety of REGN3918 in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH) Who Are Complement Inhibitor-Naive or Have Not Recently Received Complement Inhibitor Therapy
Brief Title: Study to Evaluate the Efficacy and Safety of REGN3918 in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R3918-PNH-1852; 2018-002734-20 (EudraCT Number)
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REGN3918 (Experimental): Cohort A (Dose Confirmation) If a decision is made to expand Cohort A, patients will be assigned to Cohort A.
  Cohort B (Dose Expansion) If a decision is made to progress to Cohort B, patients will be assigned to Cohort B.
  Interventions: Drug: REGN3918

INTERVENTIONS:
Drug: REGN3918 — Single intravenous (IV) dose, then a subcutaneous (SC) dose once weekly (QW).

SUMMARY:
The primary objective of the study is to demonstrate a reduction in intravascular hemolysis by REGN3918 over 26 weeks of treatment in patients with active PNH who are treatment-naive to complement inhibitor therapy or have not recently received complement inhibitor therapy.

The secondary objectives of the study are:

* To evaluate the safety and tolerability of REGN3918.
* To evaluate the effect of REGN3918 on parameters of intravascular hemolysis
* To assess the concentrations of total REGN3918 in serum.
* To evaluate the incidence of treatment-emergent anti-drug antibodies to REGN3918 over time
* To evaluate the effect of REGN3918 on patient-reported outcomes (PROs) measuring fatigue and health-related quality of life

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of paroxysmal nocturnal hemoglobinuria (PNH) confirmed by high-sensitivity flow cytometry
* PNH granulocytes > 10% at screening visit
* Active disease, as defined by the presence of 1 or more PNH-related signs or symptoms (eg, fatigue, hemoglobinuria, abdominal pain, shortness of breath [dyspnea], anemia [hemoglobin <10 g/dL], history of a MAVE [including thrombosis], dysphagia, or erectile dysfunction) or history of red blood cell (RBC) transfusion due to PNH within 3 months of screening.
* Lactate dehydrogenase (LDH) level ≥ 2 × upper limit of normal (ULN) at screening visit.

Key Exclusion Criteria:

* Prior treatment with a complement inhibitor either within 6 months prior to screening visit or at any time where the patient was refractory to complement inhibitor therapy, in the opinion of the investigator (with the exception of eculizumab refractory patients due to the C5 variant R885H/C)
* History of bone marrow transplantation
* Body weight < 40 kilograms at screening visit
* Peripheral blood absolute neutrophil count (ANC) <500/μL [<0.5 x 109/L] or peripheral blood platelet count <50,000/μL
* Documented history of systemic fungal disease or unresolved tuberculosis, or evidence of active or latent tuberculosis infection (LTBI) during screening period
* Any contraindication for receiving Neisseria meningitidis vaccination and antibiotic prophylaxis therapy as recommended in the study
* Any active, ongoing infection within 2 weeks of screening or during the screening period
* Any clinically significant abnormality identified at the time of screening that in the judgment of the Investigator or any sub-Investigator would preclude safe completion of the study or constrain endpoints assessment such as major systemic diseases, or patients with short life expectancy
* Women who are pregnant, breastfeeding, or who have a positive pregnancy test at screening visit or day 1

NOTE: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (8):
- Regeneron Study Site, Shatin, Hong Kong
- Hungary (2):
  - Regeneron Study Site, Budapest
  - Regeneron Study Site, Kaposvár
- Malaysia (3):
  - Regeneron Study Site, Kota Bharu, Kelantan
  - Regeneron Study Site, Sibu, Sarawak
  - Regeneron Study Site, Kuala Terengganu, Terengganu
- Regeneron Study Site, Seoul, South Korea
- Regeneron Study Site, Airdrie, Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency [EMA], Pharmaceuticals and Medical Devices Agency [PMDA], etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the study, the sponsor made an administrative decision to stop enrollment in order to pursue a combination program of REGN3918 & cemdisiran for treatment of Paroxysmal Nocturnal Hemoglobinuria (PNH). Study was not stopped for any safety concerns or lack of efficacy. 28 participants were screened: 4 were screen failures (1-Lost to follow-up, 1-did not meet criteria, 1-other) & 24 were enrolled & treated. Enrollment was closed at 24 participants instead of 30-42 as planned in the protocol.
Groups:
- REGN3918: Participants received a single loading dose of REGN3918 30 milligrams per kilogram (mg/kg) intravenous (IV) infusion on Day 1, followed by a maintenance regimen of 800 milligrams (mg) subcutaneous (SC) injection on Day 8 once weekly (QW) up to 26 weeks of treatment period.
Period: Overall Study
Arm/Group | REGN3918
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAF) included all enrolled participants who received any study drug.
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.4 (17.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Adequate Control of Intravascular Hemolysis
Description: Participants were considered to have had adequate control of intravascular hemolysis if all of their lactose dehydrogenase (LDH) readings from Week 4 through Week 26 inclusive had values less than or equal to ≤ 1.5 × upper limit of normal (ULN). Participants must have greater than or equal to (≥) 50 percent (%) of scheduled LDH measures in those weeks, must not have had more than (>) 2 consecutive visits without LDH measures, must not have experienced breakthrough hemolysis, and must not have discontinued study treatment early. Participants were considered not to have had adequate control of intravascular hemolysis if they failed any of these criteria.
Time Frame: Week 4 through Week 26
Population: The full analysis set (FAS) included all enrolled participants who received any study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Percentage of Participants | 75.0 [57.7 to 92.3]

2. Primary Outcome: Percentage of Participants Who Achieved Transfusion Avoidance
Description: Transfusion avoidance was defined as not having received red blood cell (RBC) transfusion during the first 26 weeks. A transfusion was counted only if it was per-protocol, that is, it followed the predefined transfusion algorithm: RBC transfusion due to a post-baseline hemoglobin level < 9 grams per deciliter (g/dL) (with anemia symptoms) or a post-baseline hemoglobin level < 7 g/dL (without anemia symptoms).
Time Frame: Up to 26 Weeks
Population: The FAS included all enrolled participants who received any study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Percentage of Participants | 87.5 [74.3 to 100.0]

3. Secondary Outcome: Percentage of Participants Who Had Breakthrough Hemolysis (BTH)
Description: Breakthrough hemolysis was defined as the measurement of LDH ≥ 2 ULN concomitant with associated signs or symptoms at any time subsequent to an initial achievement of disease control (i.e., LDH ≤ 1.5 ULN).
Time Frame: Baseline up to 26 Weeks
Population: The FAS included all enrolled participants who received any study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Percentage of Participants | 0 [0 to 0]

4. Secondary Outcome: Percentage of Participants Who Achieved Normalization of Intravascular Hemolysis
Description: A participant was considered to have achieved normalization of intravascular hemolysis if their LDH readings between Week 4 through Week 26 inclusive had values ≤ 1.0 ULN. A participant must have ≥ 50% of scheduled LDH measures in those weeks, must not have had > 2 consecutive visits without LDH measures, must not have experienced breakthrough hemolysis, and must not have discontinued study treatment early. A participant was considered not to have achieved normalization of intravascular hemolysis if they failed any of these criteria.
Time Frame: Week 4 through Week 26
Population: The FAS included all enrolled participants who received any study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Percentage of Participants | 16.7 [1.8 to 31.6]

5. Secondary Outcome: Time to First Lactate Dehydrogenase (LDH) ≤1.5 x ULN
Description: A time-to-first-event analysis was used to estimate the proportion of participants achieving transfusion avoidance at Week 26.
Time Frame: Up to Week 26
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Days | 13.625 (3.6927)

6. Secondary Outcome: Percentage of Days With LDH ≤ 1.5 ULN From Week 4 Through Week 26
Description: Percentage of days was calculated as number of days with LDH ≤ 1.5 x ULN divided by the participant's total treatment duration (total number of days on treatment from Week 4 through Week 26). LDH ≤ 1.5 x ULN was used as an indicator of adequate control of intravascular hemolysis.
Time Frame: Week 4 through Week 26
Population: The FAS included all enrolled participants who received any study drug.
Measure: Mean (Standard Deviation); unit: Percentage of Days
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Percentage of Days | 93.4 (18.76)

7. Secondary Outcome: Change From Baseline in LDH Levels at Week 26
Description: Change from baseline in LDH levels at Week 26 was reported.
Time Frame: Baseline, Week 26
Population: The FAS included all enrolled participants who received any study drug.
Measure: Least Squares Mean (Standard Error); unit: Units per liter (U/L)
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Units per liter (U/L) | -5.070 (0.1467)

8. Secondary Outcome: Percent Change From Baseline in LDH Levels at Week 26
Description: Percent change from baseline in LDH levels at Week 26 was reported.
Time Frame: Baseline, Week 26
Population: The FAS included all enrolled participants who received any study drug.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Percent Change | -81.72 (1.847)

9. Secondary Outcome: Rate of Transfusion With Red Blood Cells (RBCs)
Description: The rate of transfusion with RBCs for a participant was the total number of transfusions divided by total person-years of time on treatment.
Time Frame: Baseline up to Week 26
Population: The FAS included all enrolled participants who received any study drug.
Measure: Number (95% Confidence Interval); unit: Infusions Per Participant Year
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Infusions Per Participant Year | 1.039 [0.187 to 5.772]

10. Secondary Outcome: Number of Units of Transfusion With RBCs
Description: Transfusions with RBCs proceeded according to the following predefined criteria that triggered a transfusion; however, the actual number of units to be transfused is at the discretion of the investigator: • Transfuse with RBC(s) if the post-baseline hemoglobin level is <9 g/dL with symptoms resulting from anemia or • Transfuse with RBC(s) if the post-baseline hemoglobin level is <7 g/dL.
Time Frame: Baseline up to Week 26
Population: As per changes in planned analysis, the sponsor made an administrative decision to close enrollment for this study due to a change in the clinical development program. The sample size was determined to be too small and the decision was made to not analyze the outcome.
Measure: Mean (Standard Deviation); unit: Number of units of transfusions of RBC
Arm/Group | REGN3918
Number analyzed (Participants) | 8
Number of units of transfusions of RBC | 3.625 (4.274)

11. Secondary Outcome: Change From Baseline in RBC Hemoglobin Levels at Week 26
Description: Hemoglobin levels in participants with PNH was measured. Change from baseline in RBC hemoglobin at Week 26 was reported.
Time Frame: Baseline, Week 26
Population: The FAS included all enrolled participants who received any study drug.
Measure: Least Squares Mean (Standard Error); unit: grams per liter (g/L)
Arm/Group | REGN3918
Number analyzed (Participants) | 24
grams per liter (g/L) | 15.0 (3.24)

12. Secondary Outcome: Change From Baseline in Free Hemoglobin Levels at Week 26
Description: Change from baseline in free hemoglobin levels at Week 26 was assessed.
Time Frame: Baseline, Week 26
Population: The SAF included all enrolled participants who received any study drug. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | REGN3918
Number analyzed (Participants) | 22
milligrams per deciliter (mg/dL) | -9.19 (16.264)

13. Secondary Outcome: Change From Baseline in Total Complement Hemolytic Activity Assay (CH50) at Week 26
Description: Change from baseline in total CH50 at Week 26 was reported. Here "International units per milliliter" was abbreviated as "IU/mL".
Time Frame: Baseline, Week 26
Population: The FAS included all enrolled participants who received any study drug. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: IU/mL
Arm/Group | REGN3918
Number analyzed (Participants) | 23
IU/mL | -236.6 (0.65)

14. Secondary Outcome: Percent Change From Baseline in CH50 up to Week 26
Description: Percent change from baseline in CH50 up to Week 26 was reported.
Time Frame: Baseline up to Week 26
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | REGN3918
Number analyzed (Participants) | 23
Percent Change | -99.99 (0.243)

15. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) at Week 26
Description: The FACIT-F was a 13-item, self-reported PRO measure assessing an individual's level of fatigue during their usual daily activities over the past week. This questionnaire was part of the FACIT measurement system, a compilation of questions measuring health-related QoL in participants with cancer and other chronic illnesses. The FACIT-fatigue assessed the level of fatigue using a 4-point Likert scale ranging from 0 (not at all), 1 (a little bit), 2 (somewhat), 3 (quite a bit), 4 (very much) The sum of all responses resulted in the FACIT-F score for a total possible score of 0 to 52, with higher scores indicated greater fatigue.
Time Frame: Baseline, Week 26
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | REGN3918
Number analyzed (Participants) | 22
Score on a Scale | 9.9 (1.52)

16. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-core 30 (EORTC QLQ-C30) at Week 26
Description: The EORTC QLQ-C30 was a 30-item questionnaire used to assess symptoms and side effects of treatment and the impact on everyday life. It consists of 15 domains: 5 multi-item functioning scales (physical, role, social, emotional and cognitive), answered on a 4-point scale (1=Not at all,2=A Little,3=Quite a Bit,4=Very Much). Each score ranges from 0-100 with a higher score indicates higher level of functioning and a better QoL. A global health status/QoL scale that was answered on a 7-point scale (1=Very Poor to 7=Excellent). Each score ranges from 0-100 with a higher score indicates a better QoL. 9 symptom scales (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Insomnia, Appetite Loss, Constipation, Diarrhea, Financial Impact), answered on a 4-point scale (1=Not at all, 2=A Little, 3=Quite a Bit, 4=Very Much). Each score ranges from 0 to 100 with a higher score indicates a higher level of symptoms, and a negative change from baseline indicates an improvement in symptoms.
Time Frame: Baseline, Week 26
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | REGN3918
Number analyzed (Participants) | 22
Score on a Scale
  Global Health status/quality: Change at Week 26 | 12.509 (3.2286)
  Physical Functioning: Change at Week 26 | 17.511 (2.6767)
  Emotional Functioning: Change at Week 26 | 14.457 (3.8645)
  Social Functioning: Change at Week 26 | 15.846 (3.8036)
  Fatigue: Change at Week 26 | -18.904 (2.9899)
  Pain: Change at Week 26 | -13.537 (3.0315)
  Dyspnea: Change at Week 26 | -15.874 (4.7953)
  Cognitive Functioning: Change at Week 26 | 9.840 (2.9710)

17. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions-3 Level (EQ-5D-3L) Index Score
Description: EQ-5D-3L was a self-administered standardized instrument for use as measure of health outcome. It comprised 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension rated on 3 levels scale: 1 (no problems), 2 (some problems), 3 (extreme problems). The summed score ranges from 5-15 with "5" corresponding to no problems and "15" to severe problems in 5 dimensions. EQ-5D index calculated by applying preference-based weights (tariffs) to scores of five health state dimensions. Index values range from -1 to 1, with 0 representing a health state equivalent to death and 1 representing perfect health. Total index EQ-5D-3L summary score was weighted with a range of -0.594 (worst) to 1.0 (best).
Time Frame: Baseline, Week 26
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | REGN3918
Number analyzed (Participants) | 22
Score on a Scale | 0.136 (0.0238)

18. Secondary Outcome: Change From Baseline in EQ-5D-3L Visual Analogue Scale (VAS) at Week 26
Description: The EQ-5D-3L was a standardized instrument for use as a measure of health outcome and was administered to all participants to assess the effect of the treatment on the participants' quality of life. The EQ-5D-3L includes a visual analog scale (VAS) which is a vertical scale with numbers ranging from 0 to 100. Participants were asked to draw a line to the place on the scale that best represented how good or bad his health was on that day. The worst state a participant can imagine was marked zero, and the best state the participant can imagine was marked 100. Mean change in VAS score from baseline was reported.
Time Frame: Baseline, Week 26
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | REGN3918
Number analyzed (Participants) | 22
Score on a Scale | 8.4 (2.18)

19. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. TEAEs was defined as AEs that developed or worsened during the on-treatment period. SAE was defined as any untoward medical occurrence that resulted in any of following outcomes: death, life-threatening, required initial/prolonged in-participant hospitalization, persistent/significant disability/incapacity, congenital anomaly/birth defect/considered as medically important event. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Week 26
Population: The SAF included all enrolled participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Participants
  Participants with TEAEs | 21
  Participants with Serious TEAEs | 0

20. Secondary Outcome: Number of Participants With TEAEs Based on Severity
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. Severity of AEs was graded according to the following scale, Mild: event that does not generally interfere with usual activities of daily living; Moderate: event that interferes with usual activities of daily living, causing discomfort, permanent risk of harm; Severe: AE that interrupts usual activities of daily living, significantly affects clinical status, or may require intensive therapeutic intervention.
Time Frame: Baseline up to Week 26
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Participants
  Participants with Mild TEAEs | 13
  Participants with Moderate TEAEs | 6
  Participants with Severe TEAEs | 2

21. Secondary Outcome: Number of Participants With Clinically Meaningful Changes in Clinical Laboratory Parameters
Description: Clinical laboratory parameters included biochemistry, hematology and urinalysis. Number of participants with potential clinically significant changes in laboratory parameters which were deemed clinically meaningful by the investigator were reported.
Time Frame: Baseline up to Week 26
Population: The SAF included all enrolled participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Participants
  Hematology | 13
  Chemistry | 17
  Urinalysis | 0

22. Secondary Outcome: Number of Participants With Clinically Meaningful Changes in Vital Signs
Description: Vital sign assessments included pulse rate, blood pressure (systolic and diastolic blood pressure) and body temperature. Number of participants with potential clinically meaningful changes in vital signs which were deemed clinically significant by the investigator were reported.
Time Frame: Baseline up to Week 26
Population: The SAF included all enrolled participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Participants | 12

23. Secondary Outcome: Number of Participants With Clinically Meaningful Changes in 12-lead Electrocardiograms (ECGs)
Description: 12-lead ECGs were evaluated. Any change in ECG assessments which are deemed clinically meaningful by the investigator were reported.
Time Frame: Baseline up to Week 26
Population: The SAF included all enrolled participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Participants | 0

24. Secondary Outcome: Serum Concentrations of Total REGN3918
Description: Serum Concentrations of total REGN3918 was reported.
Time Frame: Pre-dose (Day 0), End of infusion at Days 0, 2, 7, 28, 56, 84, 112, 140, and 182
Population: The pharmacokinetic (PK) analysis set includes all participants who received any study drug and who had at least 1 non-missing result for concentration of REGN3918 following the first dose of study drug. Participants will be analyzed according to the treatment actually received. Here, "Number analyzed" signifies those participants who were evaluable at the specified time points.
Measure: Mean (Standard Deviation); unit: Milligram/liter (mg/L)
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Milligram/liter (mg/L)
  At Day 0 (Pre-dose) | 0 (0)
  At Day 0 (End of Infusion) | 605 (214)
  At Day 2 (End of Infusion) | 429 (159)
  At Day 7 (End of Infusion) | 292 (80.5)
  At Day 28 (End of Infusion): number analyzed (Participants) | 23
  At Day 28 (End of Infusion) | 324 (97.5)
  At Day 56 (End of Infusion): number analyzed (Participants) | 22
  At Day 56 (End of Infusion) | 368 (148)
  At Day 84 (End of Infusion): number analyzed (Participants) | 22
  At Day 84 (End of Infusion) | 363 (152)
  At Day 112 (End of Infusion): number analyzed (Participants) | 23
  At Day 112 (End of Infusion) | 379 (186)
  At Day 140 (End of Infusion): number analyzed (Participants) | 23
  At Day 140 (End of Infusion) | 430 (225)
  At Day 182 (End of Infusion) | 435 (221)

25. Secondary Outcome: Number of Participants With Treatment-emergent Anti-Drug Antibodies (ADA) Response to REGN3918
Description: Number of Participants with treatment-emergent ADA response to REGN3918 was reported.
Time Frame: Baseline up to Week 26
Population: The ADA analysis set (AAS) included all participants who received any study drug and who had at least 1 non-missing ADA result from the REGN3918 ADA assay after the first dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | REGN3918
Number analyzed (Participants) | 24
Participants | 0

ADVERSE EVENTS:
Time Frame: From first dose to Week 26
Arm/Group | REGN3918
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 13/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REGN3918 (N=24)
Headache (Nervous system disorders) | 9 (10)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (3)
Injection site reaction (General disorders) | 3 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/48/NCT03946748/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT03946748/SAP_001.pdf